CLINICAL TRIAL: NCT04759261
Title: SMAD4 Methylation and Expression Levels in Non-melanocytic Skin Cancers; SMAD4 Protein Positivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Metin Budak, Asist. Prof. Dr., Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/55; SMAD4 (Other: Trakya University)
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal Cell Carcinoma; Squamose Cell Carcinoma; Actinic Keratoses; SMAD4 methylation; SMAD4 expression
MeSH Terms: conditions — Carcinoma, Basal Cell; Keratosis, Actinic | interventions — Methylation

STUDY DESIGN:
Intervention Model Description: Differantiation of tumor tissues than normal tissues in same patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other)
  Interventions: Other: SMAD4 expression and methylation

INTERVENTIONS:
Other: SMAD4 expression and methylation — Effect of SMAD4 methylations on smad4 expression

SUMMARY:
Non-melanocytic skin cancers are the most common type of cancer worldwide. In the development of this cancer type, environmental factors such as UV and smoking are emphasized.

Epigenetics are genetic conditions that develop due to environmental factors and can be inherited. Epigenetic modifications such as DNA methylation play an integral role in carcinogenesis, cancer progression and metastasis.

The TGF-/ SMAD4 pathway plays a tumor suppressive role in cancer pathogenesis. Epigenetic changes in this pathway also lead to a decrease in expression level, leading to different types of cancer. However, there is no study showing the epigenetic relationship between non-melanocytic skin cancer and SMAD4 methylation.

In this study we planned, it was aimed to show the change in SMAD4 methylation and SMAD4 RNA expression level in cancerous tissue. In addition, it is planned to measure the SMAD4 protein positivity rate in non-melanocytic cancers as an immunohistochemical marker.

In this context, 60 patients who applied to Trakya University Dermatology and Venereal Diseases Outpatient Clinic and diagnosed with non-melanocytic skin cancer clinically and dermoscopically will be included in the study. Tissue materials obtained from both cancerous and intact skin of the patients will be examined in Trakya University Medical Biophysics and Medicine Pathology laboratories through various steps.

Our project is the first study to be conducted on this subject in terms of handling all non-melanocytic skin cancers, using human tissue and having a large sample.

In addition, with the data to be obtained; We think that better clarification of the role of SMAD4 in non-melanocytic cancers and the use of SMAD4 as both a prognostic factor and an immunohistochemical marker in future studies will prevent this study.

Again, we anticipate that different treatment modalities will be developed and different functional studies can be designed through this pathway.

ELIGIBILITY:
Inclusion Criteria:

1. People diagnosed clinically and dermoscopically with non-melanocytic skin cancer
2. No other cancer history
3. over 18 years old
4. Newly diagnosed
5. No systemic or topical therapy

Exclusion Criteria:

1. Under 18 and pregnant
2. People with non-melanocytic skin cancer who are in the process of follow-up and treatment
3. has another cancer history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of SMAD4 methylations and expression | 2 years
  Detection of SMAD4 methylations on tumor tissues

CONTACTS AND LOCATIONS:
Overall Officials: Metin Budak, Principal Investigator — Trakya University; Fatma El Usturali Keskin, MD, Principal Investigator — Trakya University; Yildiz Gursel, MD, Study Director — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

REFERENCES:
- [Derived] Gursel Urun Y, Budak M, Usturali Keskin E. Methylation status, mRNA and protein expression of the SMAD4 gene in patients with non-melanocytic skin cancers. Mol Biol Rep. 2023 Sep;50(9):7295-7304. doi: 10.1007/s11033-023-08656-2. Epub 2023 Jul 10. PMID 37428273